CLINICAL TRIAL: NCT06290466
Title: A Phase I, Single-center, Randomized, Double-blind, Placebo-controlled Design to Evaluate the Pharmacokinetics and Effects on QT Interval of a Single Oral Dose of FCN-437c Capsule in Healthy Subjects.
Brief Title: Clinical Study on Pharmacokinetics of FCN-437c Capsule and Its Effect on QT Interval in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ahon Pharmaceutical Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FCN-437c-CP-004
Record Dates: First submitted 2024-02-18; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Advanced Breast Cancer
Keywords: QT interval
MeSH Terms: interventions — Population Groups; FCN-437c

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FCN-437c capsule (Experimental): fasting oral, single dose.Specification :100mg
  Interventions: Drug: Low dose group; Drug: High dose group
- FCN-437c capsule Placebo (Placebo Comparator): fasting oral,single dose.Specification :100mg
  Interventions: Drug: Low dose group; Drug: High dose group

INTERVENTIONS:
Drug: Low dose group — 300 mg,single dose.
  Other Names: FCN-437c capsule or FCN-437c capsule Placebo
Drug: High dose group — 400 mg, single dose.
  Other Names: FCN-437c capsule or FCN-437c capsule Placebo

SUMMARY:
This is a single-center, randomized, double-blind, placebo-controlled Phase I clinical trial in healthy subjects.In healthy subjects, 300mg and 400mg FCN-437c capsules were taken orally for a single time. C-QTc effect model was used to evaluate the influence of blood concentration on QT interval, and the pharmacokinetic characteristics and safety of FCN-437c were also evaluated.Based on the C-QTc effect model, this study quantitatively analyzed the relationship between ΔΔQTcF and blood concentration, and evaluated the upper limit of 90% bilateral confidence interval of ΔΔQTcF corresponding to the geometric mean of Cmax at clinically relevant dose of FCN-437c capsule.

This study plans to set up 2 dose groups, low-dose group 300mg and high-dose group 400mg.Nine healthy subjects were planned to be enrolled in each dose group, with a 2:1 ratio of placebo control.

This study was carried out in the order of dose from low to high. After the administration of the low-dose group (300mg) and the safety assessment on the fourth day after administration, the study of the high-dose group (400mg) was decided through comprehensive evaluation.

ELIGIBILITY:
Inclusion Criteria:

1．Healthy adult male and female subjects (not less than 1/3 of either sex); 2．18~45 years old (including boundary values)After bilateral oophorectomy; 3．The body mass index (BMI) should be between 19.0 and 26.0 kg/m2 (including boundary values), and the weight of male subjects should not be less than 50 kg and that of female subjects should not be less than 45 kg; 4．Voluntarily sign informed consent 5．The subjects were able to communicate well with the investigators and complete the test according to protocol.

Exclusion Criteria:

Patients who meet any of the following conditions are not allowed to enter this clinical study：

1. After a comprehensive physical examination, vital signs, laboratory examination (blood routine, blood biochemistry, coagulation function, urine routine) and other abnormalities and clinical significance;
2. Hyperkalemia, hypokalemia, hypermagnesia, hypomagnesemia, hypercalcemia or hypocalcemia, which is abnormal and clinically significant as determined by the investigator;
3. Abnormal 12-lead ECG results were clinically significant, QTcF≥450 ms, PR interval ≥200 ms;QRS group duration ≥120ms;
4. Hepatitis B surface antigen or hepatitis B core antibody, hepatitis C antibody, HIV antibody or syphilis antibody positive;
5. Any drug that inhibits or induces liver drug metabolism enzymes has been used within 30 days prior to the screening period
6. Use any drug known to prolong the QT interval within 30 days prior to the screening period
7. Use of any prescription, over-the-counter, herbal or food supplements, such as vitamins and calcium supplements, in the 14 days prior to the screening period;
8. A history of any clinically serious medical conditions or conditions that the investigator believes may affect the results of the study, including but not limited to circulatory, respiratory, endocrine, nervous, digestive, urinary, or blood, immune, psychiatric, or metabolic disorders;
9. Have any conditions that may affect drug absorption, such as gastrectomy, cholecystectomy, gastric bypass, duodenotomy, colectomy, history of inflammatory bowel;
10. History of organic heart disease, heart failure, myocardial infarction, angina pectoris, coronary artery bypass grafting, angioplasty, stent stenting, congestive heart failure, uncontrolled hypotension, left ventricular ejection fraction lower than the lower limit of normal location, unexplained arrhythmia, ventricular tachycardia, atrioventricular block, and prolonged QT syndromeOr have symptoms of prolongation QT syndrome and a family history (as shown by genetic evidence or by a close relative who died of sudden cardiac death at a young age);
11. Patients who have undergone any surgery within 6 months prior to the screening period;
12. Allergy, such as a known history of allergy to two or more substances;Or who may be allergic to the drug or its excipients (e.g. Lactose T80, silica, sodium stearfumarate, etc.) as determined by the investigator;
13. Binge drinking or regular drinking in the 6 months preceding the screening period, i.e. drinking more than 14 units of alcohol per week (1 unit =360mL beer or 45 mL spirits with 40% alcohol or 150 mL wine);Or positive alcohol breath test results during the screening period;
14. Use of nicotine-containing products from 3 months prior to screening to the period of study participation;
15. Those who have a history of drug abuse or drug use 3 months before the screening period;Or positive urine drug test during screening;
16. Habitual users of grapefruit juice or excessive amounts of tea, coffee and/or caffeinated beverages who were unable to abstain during the trial period;
17. Patients with a history of needle fainting and blood fainting, difficulty in blood collection or inability to tolerate venous puncture blood collection
18. Participation in any other clinical trials (including drug and device trials) within 3 months prior to the screening period;
19. Those who were vaccinated within 1 month prior to screening or planned to be vaccinated during the trial period;
20. Pregnant or lactating women;
21. Participants who planned to have children or donate sperm during the study period and six months after completion of the study, or did not agree that participants and their spouses should use strict contraceptive methods during the study period and six months after completion of the study
22. Patients who had blood loss or blood donation of up to 400 mL within 3 months prior to the screening period, or received a blood transfusion within 1 month
23. Subjects with any factors deemed unsuitable for participation in the study by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2023-02-08 (Actual); Study Completion 2023-02-08 (Actual)

PRIMARY OUTCOMES:
ΔΔQTcF | 2hours before administration and 48hours and 192hours after administration
  The Cmax geometric mean corresponds to the upper 90% bilateral confidence interval of ΔΔQTcF

SECONDARY OUTCOMES:
adverse events | Trial period to day 21 after administration
  The number, frequency and incidence of adverse events
Physical examination | From 1 day before administration to 21 days after administration
  Descriptive statistics on physical examination indicators visited and their changes from baseline
Axillary temperature | From 2.0 hours before administration to 21 days after administration
  Descriptive statistics of vital signs at each visit and their change from baseline
blood pressure | From 2.0 hours before administration to 21 days after administration
  Descriptive statistics of vital signs at each visit and their change from baseline
pulse | From 2.0 hours before administration to 21 days after administration
  Descriptive statistics of vital signs at each visit and their change from baseline
Ecg monitoring and electrocardiogram | Trial period to day 21 after administration
  QTcF
laboratory examination | Trial period to day 21 after administration
  Descriptive statistics were collected for each laboratory indicator visited and its change from baseline
Plasma concentration and pharmacokinetic parameters | 60 minutes before dosing to day 9 after dosing
  Cmax
Plasma concentration and pharmacokinetic parameters | 60 minutes before dosing to day 9 after dosing
  AUC0-t
Plasma concentration and pharmacokinetic parameters | 60 minutes before dosing to day 9 after dosing
  AUC0-∞
Plasma concentration and pharmacokinetic parameters | 60 minutes before dosing to day 9 after dosing
  Tmax
Plasma concentration and pharmacokinetic parameters | 60 minutes before dosing to day 9 after dosing
  T1/2
Plasma concentration and pharmacokinetic parameters | 60 minutes before dosing to day 9 after dosing
  CL/F
Plasma concentration and pharmacokinetic parameters | 60 minutes before dosing to day 9 after dosing
  VZ/F
Plasma concentration and pharmacokinetic parameters | 60 minutes before dosing to day 9 after dosing
  MRT
Plasma concentration and pharmacokinetic parameters | 60 minutes before dosing to day 9 after dosing
  AUC_%Extrap

CONTACTS AND LOCATIONS:
Overall Officials: Haiyan Li, MD, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zhao L, Sun Y, Yang X, Tian L, Li L, Wang F, Niu X, Diao L, Li H. No QTc prolongation with CDK 4/6 inhibitor FCN-437c: results of a concentration-QTc analysis from a dedicated study in adult healthy subjects. Front Pharmacol. 2024 Aug 12;15:1433663. doi: 10.3389/fphar.2024.1433663. eCollection 2024. PMID 39188943